CLINICAL TRIAL: NCT07335874
Title: Overview of Targeted Screening for Congenital Infection Guided by Neonatal Hearing Screening
Acronym: cCMV-DNS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9689
Record Dates: First submitted 2026-01-02; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Neonatal Hearing Loss
Keywords: Neonatal hearing loss; Cytomegalovirus infection; Congenital infection; Sensorineural hearing loss
MeSH Terms: conditions — Cytomegalovirus Infections; Hearing Loss, Sensorineural

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cytomegalovirus (CMV) infection is the most common congenital infection. It is the second leading cause of sensorineural hearing loss after genetic causes and the leading cause of motor delay. It can also cause ophthalmological or biological abnormalities (hepatic cytolysis, thrombocytopenia, etc.). Currently, routine screening during pregnancy or at birth is not recommended.

90% of infected infants are asymptomatic at birth. However, 10 to 25% of them present with hearing loss at birth or will develop it in their first years of life. This hearing loss is progressive.

In the context of deafness, detecting congenital CMV infection helps explain the cause of hearing loss (a recurring question from parents) and allows for tailored management and follow-up (progressive deafness, bilateral involvement). Its detection also enables appropriate pediatric monitoring (neurological, ophthalmological, etc.). Screening for congenital CMV infection (cCMV), guided by neonatal hearing screening, has been recommended by the French High Council for Public Health (HCSP) since 2018.

In cases of confirmed congenital CMV infection, an ophthalmological examination (fundus examination), hearing test, brain imaging, and blood tests are performed.

The investigators wish to collect data from targeted screening for congenital CMV infection at the Strasbourg University Hospitals (HUS) to ensure comprehensiveness and to study CMV-related conditions in these screened children.

ELIGIBILITY:
Inclusion Criteria:

* Minors aged 0 to 1 month at the time of newborn hearing screening
* Subject with inconclusive newborn hearing screening (NHS) on unilateral or bilateral T2 (inconclusive retest) between August 2024 and the end of July 2025.

Exclusion Criteria:

* Positive CMV PCR after 1 month of life
* CMV PCR performed for another indication.

Ages: 0 Years to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: - Minors aged 0 to 1 month at the time of newborn hearing screening with inconclusive newborn hearing screening (NHS) on unilateral or bilateral T2 (inconclusive retest) between August 2024 and the end of July 2025.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06-16 (Estimated)

PRIMARY OUTCOMES:
CMV PCR rates (in %) in infants with inconclusive T2 at the newborn hearing screening (DNS) | Up to 12 months
  CMV PCR rates in infants with inconclusive T2 at the newborn hearing screening (DNS) (number of PCR tests performed / total number of infants with inconclusive T2)

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'ORL et de Chirurgie Cervico-faciale - CHU de Strasbourg - France, Strasbourg, France